CLINICAL TRIAL: NCT04122274
Title: Comparing and Interactive Concussion Education Platform to Current Education Standards: A Randomized Control Trial
Brief Title: Comparing and Interactive Concussion Education Platform to Current Education Standards
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 19-1633
Record Dates: First submitted 2019-10-08; First posted 2019-10-10 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-04

CONDITIONS: Concussion, Brain
Keywords: Concussion, Education
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education Sheet and Sham Intervention (Sham Comparator): Participants will be asked to fill out a pre-intervention survey to assess existing concussion knowledge, perceived norms, attitudes, and behavioral intentions. Afterward, the NCAA concussion education fact sheet will be viewed along with the viewing of the sham intervention. Following the intervention, a post-intervention survey re-assessing the constructs from the pre-intervention survey will be completed. May be completed in-person or virtually.
  Interventions: Behavioral: NCAA education sheet; Behavioral: Decision-based interactive concussive education platform
- Education Sheet and Decision-based interactive intervention (Experimental): Participants will be asked to fill out a pre-intervention survey to assess existing concussion knowledge, perceived norms, attitudes, and behavioral intentions. Afterward, the NCAA concussion education fact sheet will be viewed along with the viewing of a decision- based interactive concussion education platform intervention. Following the intervention, a post-intervention survey re-assessing the constructs from the pre-intervention survey will be completed. May be completed in-person or virtually.
  Interventions: Behavioral: NCAA education sheet; Behavioral: Sham Intervention

INTERVENTIONS:
Behavioral: NCAA education sheet — A fact sheet that includes information about basic signs and symptoms of a concussion as well as steps to take if an individual sustains a concussion and reinforces the need to report the injury.
Behavioral: Sham Intervention — An approximately 7-minute video that includes information about basic sports nutrition facts.
  Arms: Education Sheet and Decision-based interactive intervention
Behavioral: Decision-based interactive concussive education platform — A platform grounded in theoretical frameworks including the socioecological model and theory of planned behavior. It includes a short video to provide an overview of key lessons, a short quiz, and additional resource links that conclude the module.
  Arms: Education Sheet and Sham Intervention

SUMMARY:
Purpose: The purpose of this study is to evaluate the effectiveness of a theory- driven education platform to improve concussion-related norms and perceptions in an effort to improve student-athletes concussion-related decision-making.

Participants: 80 college-aged recreational athletes.

Procedures: The study is a single-blind (participants) randomized control trial where participants will complete a previously validated survey assessing concussion knowledge, perceived norms, attitudes, and behavioral intentions immediately pre- and post-receipt of their designated intervention. Participants will also complete the previously validated survey two-week post receipt of their designated intervention. The interventions include an interactive concussion education platform along with the NCAA (National Collegiate Athletic Association) concussion education sheet and the NCAA concussion education sheet alone (with a sham educational intervention similar in length to the concussion education platform).

DETAILED DESCRIPTION:
A convenience sample of participants will be recruited from the University of North Carolina at Chapel Hill student-body from November-January via campus emails, in-class recruitment, flyers/informational sheets, and word of mouth from fellow participants. During the beginning of recruitment, efforts were targeted towards males with participant numbers being carefully monitored. Recruitment will be targeted to recruit an even number of males and females. Interested participants will be contacted to confirm interest and those who remained interested will be scheduled to complete the study session. Participants will report to an on-campus athletic training facility or research laboratory or may report/complete study activities virtually.

Participants will then complete the written, informed consent process. The consent form indicated that they would be completing a sport-related educational intervention to not disclose the information they would receive and to keep participants blind to their intervention group assignment. Participants will not be explicitly told that it is a study evaluating concussion education, but rather an injury and nutrition study, to reduce bias. Once the consent form was signed, participants were assigned a unique identifier and randomized (simple) without replacement to one of the two study arms, using a pre-determined random number generator in Excel. Participants then completed the pre- questionnaire in a quiet location via a tablet/computer provided by the research team or virtually. There was no time limit for completion of the questionnaire. The survey will feature an item that prompts individuals if they miss a question, but does not force participants to respond. After initial questionnaire completion, participants completed their assigned intervention (decision-based interactive concussion education platform + NCAA concussion education sheet versus NCAA education sheet). Immediately following their respective intervention, athletes completed the questionnaire again. Upon completing the post-intervention questionnaire, the participant's participation in the study is complete and they will receive an incentive. Following each survey, a research team member will verify and assess for missing answers, allowing participants to complete any missed questions that they wish to answer. Two weeks following the post-intervention survey, participants will be contacted again to complete the same questionnaire to assess retention of concussion knowledge, perceived norms, attitudes, and behavioral intentions. At this two-week post time point, participants will be informed of the true purpose of the study and be provided access to the BANK (Behaviors, Attitudes, Norms, and Knowledge) platform.

ELIGIBILITY:
Inclusion Criteria:

* Rostered club sport and/or recreational athletes at a single institution will be recruited for participation in this study.

Exclusion Criteria:

* There are no additional exclusion criteria for rostered club and intramural athletes at the study institution

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2019-10-21 (Actual); Primary Completion 2022-04-21 (Actual); Study Completion 2022-04-21 (Actual)

PRIMARY OUTCOMES:
Perceived Behavioral Norms Change Score | From pre to post intervention, an approximate total of up to thirty minutes.
  Participants are asked seven questions on a previously validated BANK survey identifying what an athlete thinks are important to people in his or her environment would do with respect to concussion reporting. Each item is added together to compute an overall perceived behavioral norms score. The difference between the intervention and post-intervention total score is calculated to compute a change score.Scoring scale ranges from a minimum of 7 to a maximum of 49, where higher scores indicate more favorable perceived norms.
Behavioral Intention Change Score | From pre to post intervention, an approximate total of up to thirty minutes.
  Participants are asked a three questions on a previously validated BANK survey assessing intention to disclose a concussion or concussion-like symptoms. The items are totaled to compute an overall behavioral intention score. The difference between the pre-intervention and post-intervention score is calculated to compute a change score.Scoring scale ranges from a minimum of 3 to a maximum of 21, where a higher score indicates a better likelihood that an individual will disclose concussion-like symptoms.

SECONDARY OUTCOMES:
Pre-Intervention Concussion Knowledge Score | Within approximately 15 minutes prior to viewing intervention
  Participants are asked thirty-nine questions on a previously validated BANK survey concerning information. regarding signs & symptoms, diagnosis, treatment, and return to play following a sport-related concussion. Each item is added together to compute an overall concussion knowledge score. Scoring scale ranges from a minimum of 0 to a maximum 39, where a higher score indicated better concussion knowledge.
Pre-intervention Perceived Behavioral Norms Score | Within approximately 15 minutes prior to viewing intervention
  Participants are asked seven questions on a previously validated BANK survey identifying what an athlete thinks are important to people in his or her environment would do with respect to concussion reporting. Each item is added together to compute an overall perceived behavioral norms score. Scoring scale ranges from a minimum of 7 to a maximum 49, where high scores indicate more favorable perceived norms.
Pre-Intervention Attitudes Score | Within approximately 15 minutes prior to viewing intervention
  Participants are asked six survey items identifying an individual's beliefs about a certain behavior (e.g., concussion disclosure).Each item is added together to compute an overall attitude score. Scoring scale ranges from a minimum of 6 to a maximum of 42, where higher scores indicate more favorable attitudes.
Pre-Intervention Behavioral Intention Score | Within approximately 15 minutes prior to viewing intervention
  Participants are asked three questions on a previously validated BANK survey assessing intention to disclose a concussion or concussion-like symptoms. The items are totaled to compute an overall behavioral intention score. Scoring scale ranges from a minimum of 3 to a maximum of 21, where a higher score indicates a better likelihood to disclose concussion-like symptoms.
Post-Intervention Concussion Knowledge Score | Up to approximately 30 minutes after viewing intervention
  Participants are asked thirty-nine questions on a previously validated BANK survey concerning information regarding signs & symptoms, diagnosis, treatment, and return to play following a sport-related concussion. Each item is added together to compute an overall knowledge score. The scoring scale ranges from a minimum of 0 to a maximum of 39, where a higher score indicates better concussion knowledge.
Post-intervention Perceived Behavioral Norms Score | Up to approximately 30 minutes after viewing intervention
  Participants are asked seven questions on a previously validated BANK survey identifying what an athlete thinks are important to people in his or her environment would do with respect to concussion reporting. Each item is added together to compute an overall perceived behavioral norms score. Scoring scale ranges from a minimum of 7 to a maximum of 49, where a higher score indicates more favorable perceived norms.
Post-Intervention Attitudes Score | Up to approximately 30 minutes after viewing intervention
  Participants are asked six survey items identifying an individual's beliefs about a certain behavior (e.g., concussion disclosure). Each item is added together to compute an overall attitude score. Scoring scale ranges from a minimum of 6 to a maximum of 42, where a higher score indicates more favorable attitudes.
Post-Intervention Behavioral Intention Score | Up to approximately 30 minutes after viewing intervention
  Participants are asked three questions on a previously validated BANK survey assessing intention to disclose a concussion or concussion-like symptoms. The items are totaled to compute an overall behavioral intention score. The scoring scale ranges from a minimum of 3 to a maximum of 21, where a higher score indicates a better likelihood that the individual will disclose concussion-like symptoms.
Concussion Knowledge Change Score | From pre to post intervention, an approximate total of up to thirty minutes.
  Participants are asked thirty-nine questions on a previously validated BANK survey concerning information. regarding signs & symptoms, diagnosis, treatment, and return to play following a sport-related concussion. Each item is added together to compute an overall knowledge score. The difference between the pre-intervention and post-intervention total score is calculated to compute a change score. Scoring scale ranges from a minimum of 0 to a maximum of 39, where higher scores indicate better concussion knowledge.
Attitudes Change Score | From pre to post intervention, an approximate total of up to thirty minutes.
  Participants are asked six survey items identifying an individual's beliefs about a certain behavior (e.g., concussion disclosure). Each item is added together to compute an overall attitude score. The difference between the pre-intervention and post-intervention total score is calculated to compute a change score. Scoring scale ranges from a minimum of 6 to a maximum of 42, where higher scores indicate more favorable attitudes.
Concussion Knowledge Retention Score | Within approximately 2 weeks following the viewing of the intervention
  Participants are asked thirty-nine questions on a previously validated BANK survey concerning information. regarding signs & symptoms, diagnosis, treatment, and return to play following a sport-related concussion. Each item is added together to compute an overall knowledge score. The scoring scale ranges from a minimum of 0 to a maximum of 39, where higher scores indicate better concussion knowledge.
Perceived Behavioral Norms Retention Score | Within approximately 2 weeks following the viewing of the intervention
  Participants are asked seven questions on a previously validated BANK survey identifying what an athlete thinks are important to people in his or her environment would do with respect to concussion reporting. Each item is added together to compute an overall perceived behavioral norms score. Scoring scale ranges from a minimum of 7 to a maximum of 49, where higher schools indicate more positive perceived norms.
Attitudes Retention Score | Within approximately 2 weeks following the viewing of the intervention
  Participants are asked six survey items identifying an individual's beliefs about a certain behavior (e.g., concussion disclosure). Each item is added together to compute an overall attitude score. The scoring scale ranges from a minimum of 6 to a maximum of 42, where higher scores indicate more favorable attitudes.
Behavioral Intention Retention Score | Within approximately 2 weeks following the viewing of the intervention
  Participants are asked three questions on a previously validated BANK survey assessing intention to disclose a concussion or concussion-like symptoms. The items are totaled to compute an overall behavioral intention score. The scoring scale ranges from a minimum of 3 to a maximum 21, where a higher score indicates a better likelihood that an individual will disclose concussion-like symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Johna K Register-Mihalik, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, SAP
Time Frame: 9 to 36 months following publication
Access Criteria: IRB, IEC, or REB and an executed data use/sharing agreement with the University of North Carolina at Chapel Hill